CLINICAL TRIAL: NCT06149195
Title: 18F-meta-fluorobenzylguanidine Cardiac Imaging for Evaluation of Chronic Heart Failure
Brief Title: 18F-MFBG Cardiac Imaging for Heart Failure Administration
Status: Enrolling by invitation | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Associate senior physician, Sichuan Provincial People's Hospital
Other Study IDs: CMFBG202311
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Rest Gated Myocardial Perfusion Imaging in Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- positive: positive imaging, referring to the tracer absented in the left myocardium whether diffuse or localized on 18F-FMBG cardiac imaging.
  Interventions: Diagnostic Test: Standard medical care for heart failure

INTERVENTIONS:
Diagnostic Test: Standard medical care for heart failure — Standard treatment and care for heart failure patients from the heart failure center of Sichuan Provincial People's Hospital.

SUMMARY:
The clinical feasibility of 18F-FMBG cardiac PET imaging will be observed in sympathetic nervous system activity in patients with heart failure, predicted cardiac events, guided ICD implantation, and evaluated therapy efficiency.

DETAILED DESCRIPTION:
This is a prospective, single-center clinical study, using18F-meta-fluorobenzylguanidine (18F-MFBG) cardiac PET imaging to present the sympathetic nerve status in heart failure, including ICD implantation. Through follow-up, we analyze the correlation between the distribution of the tracer in the heart and the functions and progression of the patients, including the occurrence of ventricular arrhythmias and sudden cardiac death, And further investigate the guiding value of 18F-MFBG cardiac sympathetic nerve imaging in the screening of ICD implantation patients, including primary and secondary prevention, reducing the cost of ICD implantation and related complications. Furthermore, to evaluate the therapy efficacy for these patients with heart failure using 18F-MFBG cardiac imaging has been considered.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinically confirmed patient with chronic heart failure, LVEF ≤ 40%, cardiac function NYHA 2-3 grade, survival period greater than 1 year, evaluated by the Heart Failure Center of Sichuan Provincial People's Hospital.
* 2. Chronic heart failure patients were evaluated by the Cardiology Department of Sichuan Provincial People's Hospital 5-10 days before ICD implantation.
* 3. All patients above have signed an informed consent form.

Exclusion Criteria:

* 1. Heart failure, heart function NYHA levels ⅠOR Ⅳ.
* 2. The patient has already implanted ICD or CRT.
* 3. Heart transplant patients.
* 4. Patients with malignant tumors.
* 5. Heart valve disease.
* 6. Myocardial infarction occurred within the past three months.
* 7. The patient has contraindications for ICD implantation surgery.
* 8. The patient does not cooperate or is unwilling to conduct the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: enrolling patients with chronic heart failure with a heart function of NYHA Class II-III.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
observe the 18F-MFBG distribution of the myocardium in heart failure patients | 1 year
  18F-MFBG PET cardiac sympathetic nerve imaging was performed after injection of 30 minutes and 3 hours. The imaging agent distribution of left ventricular walls was observed at three axis positions (short axis, horizontal long axis, and vertical long axis). Target heart maps (17 segments) were obtained using Cedars QPS software to obtain radiation distribution counts (SMSe, SMSlate).

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Ling Ding, Study Director — China, Sichuan Departments of Nuclear Medicine, Sichuan Provincial People's Hospita
Locations (1):
- Zhi Ling Ding, Chengdu, Sichuan, China